CLINICAL TRIAL: NCT04250974
Title: Single-blinded, Randomized Preliminary Study Evaluating the Effects of Electroacupuncture for Postoperative Pain Relief in Patients With Distal Radius Fracture.
Brief Title: Evaluaing the Effects of Electroacupuncture for Postoperative Pain Relief in Patients With Distal Radius Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH108-REC1-140
Record Dates: First submitted 2020-01-22; First posted 2020-01-31 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain Relief
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electroacupuncture (Experimental): electroacupuncture at points after surgery
  Interventions: Other: electroacupuncture
- electroacupuncture non-point (Sham Comparator): electroacupuncture at non-points after surgery
  Interventions: Other: electroacupuncture
- Control group (No Intervention): only oral or injection painkiller were used after surgery

INTERVENTIONS:
Other: electroacupuncture — acupuncture with electricity
  Arms: electroacupuncture; electroacupuncture non-point

SUMMARY:
Single-blinded, randomized preliminary study evaluating the effects of electroacupuncture for postoperative pain relief in patients with distal radius fracture.

Distal radius fracture is extremely common, and it is about 10% of all fractures in the human body. Therefore, the distal radius is the most frequently fractured part of the upper limbs of the human body. Once the fracture occurs, internal fixation is the main surgical procedure. The postoperative analgesic method is generally oral or injection analgesic. In recent years, electroacupuncture(EA) has been widely used to relieve pain after surgery, and many studies have confirmed that it is effective. However, there is no evaluation of analgesic efficacy after the surgery of distal radius fracture. Therefore, it is hoped that the efficacy of EA for analgesia after the surgery of distal radius fracture is demonstrated by this study. And, the investigators also hope the investigators can reduce the use of painkillers through EA.

Methods: It is expected that 30 patients will be randomly assigned to the following groups: EA group,EA at points; non-point group, EA at non-points, control group without EA

1. EA group:EA at points after surgery
2. non-point group: EA at non-points after surgery
3. Control group: no EA

DETAILED DESCRIPTION:
Single-blinded, randomized preliminary study evaluating the effects of electroacupuncture for postoperative pain relief in patients with distal radius fracture.

Distal radius fracture is extremely common, and it is about 10% of all fractures in the human body. Therefore, the distal radius is the most frequently fractured part of the upper limbs of the human body. Once the fracture occurs, internal fixation is the main surgical procedure. The postoperative analgesic method is generally oral or injection analgesic. In recent years, electroacupuncture(EA) has been widely used to relieve pain after surgery, and many studies have confirmed that it is effective. However, there is no evaluation of analgesic efficacy after the surgery of distal radius fracture. Therefore, it is hoped that the efficacy of EA for analgesia after the surgery of distal radius fracture is demonstrated by this study. And, the investigators also hope the investigators can reduce the use of painkillers through EA.

Methods: It is expected that 30 patients will be randomly assigned to the following groups: EA group,EA at points; non-point group, EA at non-points, control group without EA

1. EA group:EA at points after surgery
2. non-point group: EA at non-points after surgery
3. Control group: no EA Mode of operation: After the patient has returned to the recovery room, perfom EA, and take the needle after 30 minutes. Perform another 30 minutes after 24 hours, and then statistics.

Acupoint selection:

1. true acupoints: needles were inserted to Taichong (LR3 ) and Taixi (KI3) contralateral to the operated leg and deqi sensation elicited at acupoints
2. false point: the needles were inserted to Kunlun(BL60) and Shugu(BL65) contralateral to the operated leg and deqi sensation elicited at acupoints

Data collection:

1. Record the time required for the first injection of analgesics
2. The number of doses of oral painkiller used in 36 hours after surgery (count)
3. The number of doses of injection painkiller used in 36 hours after surgery (count)
4. Use the visual analog scale (VAS) to assess the patient's pain level

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic specialist diagnoses distal radius fracture and undergoes internal fixation
* Age between 20 and 70

Exclusion Criteria:

* Allergic to painkillers
* Have a serious heart rhythm
* epilepsy
* Severe pulmonary heart disease
* History of mental illness
* History of drug abuse
* received acupuncture treatment within 1 month

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-11-28 (Estimated); Study Completion 2020-11-28 (Estimated)

PRIMARY OUTCOMES:
the time required for the first injection of analgesics | in 36 hours after surgery
  Record the time required for the first injection of analgesics
the number of doses of injection painkiller | in 36 hours after surgery
  Record the number of doses of injection painkiller

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Cheng Chiu, MD, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, No. 2, Yude Rd, North District, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No